CLINICAL TRIAL: NCT06349954
Title: Effectiveness and Safety of Single-session Endoscopic Stone Extraction for Acute Cholangitis Associated With Choledocholithiasis
Brief Title: Effectiveness and Safety of Single-session Endoscopic Stone Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BFHHZS20240064
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-01

CONDITIONS: Choledocholithiasis With Acute Cholangitis
Keywords: Acute Cholangitis; Endoscopic Retrograde Cholangiopancreatography; Choledocholithiasis
MeSH Terms: conditions — Choledocholithiasis

STUDY DESIGN:
Intervention Model Description: All patients will be randomly allocated into single-session group or two-session group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- single-session treatment group (Experimental): single-session ERCP
  Interventions: Procedure: single-session ERCP
- two-session treatment group (Experimental): two-session ERCP
  Interventions: Procedure: two-session ERCP

INTERVENTIONS:
Procedure: single-session ERCP — directly endoscopic stone extraction
  Arms: single-session treatment group
Procedure: two-session ERCP — early endoscopic drainage followed by endoscopic stone extraction
  Arms: two-session treatment group

SUMMARY:
This is a prospective study, including approximately 64 patients with acute cholangitis accompanied with choledocholithiasis at Beijing Friendship Hospital. All patients will be randomly allocate into single-session or two-session endoscopic stone extraction. The investigators assessed the outcomes of single-session and two-session endoscopic stone extraction.

DETAILED DESCRIPTION:
Acute cholangitis is an acute inflammation caused by obstruction of the bile duct, of which choledocholithiasis is the most common cause. Without timely removal of the obstruction or control of the infection, cholangitis can get worse and even become life-threatening. Therefore, timely and effective treatment is essential for patients with acute cholangitis combined with choledocholithiasis. Endoscopic retrograde cholangiography (ERCP) is used as the first-line treatment for choledocholithiasis-associated acute cholangitis. Previous guidelines recommended two-session endoscopic therapy. Endoscopic biliary drainage as the initial treatment, followed by endoscopic stone extraction after cholangitis improved. In recent years, studies have found that single-session endoscopic stone extraction is safe and effective for patients without serious organ function impairment. Meanwhile, single-session endoscopic lithotomy can avoid the second ERCP intervention, which can relieve the pain of patients, reduce medical costs and shorten the length of hospital stay. However, there is still insufficient evidence on the effectiveness and safety of early single-session ERCP lithotomy. The aim of this study is to evaluate the efficacy and safety of single-session endoscopic stone extraction for acute cholangitis associated with choledocholithiasis, so as to provide reference of clinical treatment.

In a prospective study, approximately 64 patients with acute cholangitis accompanied with choledocholithiasis will be involved. The investigators assessed the outcomes of single-session and two-session endoscopic stone extraction.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years old and ≤90 years old
* 2. Patients met the Tokyo Guidelines 2018 (TG18) diagnosis of Grade I or Grade II acute cholangitis
* 3. Imaging examination confirmed the presence of choledocholithiasis

Exclusion Criteria:

* 1. Common bile duct with benign or malignant stenosis
* 2. Changes in the anatomical structure of the stomach or duodenum
* 3. Patients with common biliary duct or pancreatic duct stent
* 4. Patients complicated with acute pancreatitis
* 5. Patients who underwent endoscopic intervention, percutaneous transhepatic cholangio drainage (PTCD) or other invasive interventions before admission
* 6. Patients with cardiac failure, respiratory failure or consciousness disorder can not tolerate endoscopic operation
* 7. Patients who have coagulation dysfunction or are taking anticoagulation and antiplate drugs
* 8. Imaging examination showed that the maximum diameter of choledocholithiasis was more than 1.5cm

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Success rate of complete stone removal | during the operation
  Segmental angiography was performed by balloon closure to determine the presence or absence of negative stone shadow
ERCP-related complication rate | from the operation to 1 month after the operation
  The complications include pancreatitis, hemorrhage, perforation, pneumonia, etc. The results of intraoperative endoscopic observation, postoperative symptoms and signs, blood routine examination, amylase, lipase, and imaging and endoscopic examination were measured.

SECONDARY OUTCOMES:
Length of stay | perioperatively
  Total time from admission to discharge.
Hospital expenses | perioperatively
  Total expenses from admission to discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Fujing Lv, M.D., Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China